CLINICAL TRIAL: NCT00681564
Title: Impact of Periodontal Therapy on Endothelial Function
Brief Title: Periodontal Infection and Endothelial Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad del Valle, Colombia (Other)
Responsible Party: Principal Investigator, Jorge Hernán Ramírez, principal investigator, Universidad del Valle, Colombia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: COLCIENCIAS 110634319239
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Results first posted 2014-04-01 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-03

CONDITIONS: Periodontitis
Keywords: Periodontitis; Oral health; Cardiovascular disease
MeSH Terms: conditions — Periodontitis; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- One-Stage Full-Mouth Disinfection (Experimental): Scaling and root planing, four quadrants in one session Tongue brushing with a 1% chlorhexidine gel (1 minute) Mouth rinsing with a 0.2% chlorhexidine solution for (2 minutes) Subgingival chlorhexidine (1%) irrigation in all pockets Twice daily rinsing with clorhexidine (1 minute) during fourteen days after the periodontal intervention Basic oral hygiene instructions Dental extractions will be performed at the end of patient followup (only in cases of teeth that could not be saved)
  Interventions: Procedure: One-Stage Full-Mouth Disinfection
- Periodontal care (Active Comparator): Basic oral hygiene instructions Supragingival plaque removal
  Interventions: Procedure: Periodontal care

INTERVENTIONS:
Procedure: One-Stage Full-Mouth Disinfection — * Scaling and root planing, four quadrants in one session
  * Tongue brushing with a 1% chlorhexidine gel (1 minute)
  * Mouth rinsing with a 0.2% chlorhexidine solution for (2 minutes)
  * Subgingival chlorhexidine (1%) irrigation in all pockets
  * Twice daily rinsing with clorhexidine (1 minute) during fourteen days after the periodontal intervention
  * Basic oral hygiene instructions
  * Dental extractions will be performed at the end of patient followup (only in cases of teeth that could not be saved)
  Arms: One-Stage Full-Mouth Disinfection
Procedure: Periodontal care — * Basic oral hygiene instructions
  * Supragingival plaque removal
  Arms: Periodontal care

SUMMARY:
The purpose of this study is to determine the effect of periodontal therapy on endothelial function and other biomarkers of cardiovascular disease

DETAILED DESCRIPTION:
Periodontitis is one of the most prevalent chronic diseases and a frequent cause of tooth loss. Accumulation of subgingival dental biofilm in susceptible individuals is associated with an inflammatory host response characterized by the production of Matrix Metalloproteinases, reduction in collagen synthesis, increase in cytokine gene expression, and apoptosis of gingival fibroblasts. Finally, inflammation leads to destruction of periodontal ligament, alveolar bone resorption, and chronic periodontitis.

Periodontitis is associated with increased serum levels of inflammatory cytokines and acute phase reactants. Multiple case-control and cohort studies have suggested that periodontitis is an independent risk factor for cardiovascular events, diabetic end-organ damage, pregnancy complications and respiratory diseases. Recent interventional studies have found that periodontal therapy could increase endothelium-dependent brachial artery flow-mediated dilation.

The purpose of this controlled clinical trial is to determine the effect of periodontal therapy on endothelial function in subjects with moderate to severe chronic periodontitis. Furthermore, the relationship between putative periodontal pathogens and endothelial function will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 25 years of age or older
* Three or more periodontal pockets with a probing depth (PD) > 5mm
* Have at least 20 natural teeth
* Provide informed consent and willingness to cooperate with the study protocol

Exclusion Criteria:

* History of antibiotic use in the previous three months
* Pregnant or lactating females
* Treatment with antihypertensive, antilipemic, antiarrhythmic, and other cardiovascular drugs
* Systemic diseases such as diabetes, HIV/AIDS, liver disease, chronic renal failure, tuberculosis, and autoimmune diseases
* Previous history of cardiovascular disease: Acute myocardial infarct, stable angina, unstable angina, heart failure, atrial fibrillation, atrioventricular block, peripheral vascular disease, cerebrovascular accident
* Patients who received periodontal treatment within the last 3 months
* Patients who require antibiotic prophylaxis before examination or treatment
* Patients with mental retardation and dementia

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2008-05; Primary Completion 2011-03 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo Contreras, DDS, MS, PhD, Principal Investigator — Universidad del Valle; Jorge H Ramirez, MD, MS, Principal Investigator — Universidad del Valle
Locations (2):
- Colombia (2):
  - Red de Salud de Ladera E.S.E. Servicio de Odontología, Cali, Valle del Cauca Department
  - Universidad del Valle, Facultad de Salud, Escuela de Odontología, Cali, Valle del Cauca Department

REFERENCES:
- [Result] Ramirez JH, Parra B, Gutierrez S, Arce RM, Jaramillo A, Ariza Y, Contreras A. Biomarkers of cardiovascular disease are increased in untreated chronic periodontitis: a case control study. Aust Dent J. 2014 Mar;59(1):29-36. doi: 10.1111/adj.12139. Epub 2014 Feb 4. PMID 24495202
- [Derived] Ramirez JH, Arce RM, Contreras A. Periodontal treatment effects on endothelial function and cardiovascular disease biomarkers in subjects with chronic periodontitis: protocol for a randomized clinical trial. Trials. 2011 Feb 16;12:46. doi: 10.1186/1745-6215-12-46. PMID 21324167

RESULTS

PARTICIPANT FLOW:
Recruitment Details: rom April 2008 to March 2011 three hundred and six subjects were assessed for eligibility to participate in this randomized clinical trial. One hundred and two patients were randomized to the control (n=55) and treatment group (n=47). At 12 weeks of follow-up, 47 patients (control group) and 41 patients (treatment group) completed the study.
Pre-assignment Details: Two hundred and four patients were excluded from this study for the following reasons: no fulfillment of inclusion criteria (n=183), refusal to participate (n=4), not assistance to study appointments (n=15), and another reasons (n=2).
Groups:
- Periodontal Intervention (Experimental): One-Stage Full-Mouth Disinfection: - Scaling and root planing, four quadrants in one session
  * Tongue brushing with a 1% chlorhexidine gel (1 minute)
  * Mouth rinsing with a 0.2% chlorhexidine solution for (2 minutes)
  * Subgingival chlorhexidine (1%) irrigation in all pockets
  * Twice daily rinsing with clorhexidine (1 minute) during fourteen days after the periodontal intervention
  * Basic oral hygiene instructions
  * Dental extractions will be performed at the end of patient followup (only in cases of teeth that could not be saved)
- Periodontal Prophylaxis (Active Comparator): Periodontal care: - Basic oral hygiene instructions
  - Supragingival plaque removal
Period: Overall Study
Arm/Group | Periodontal Intervention (Experimental) | Periodontal Prophylaxis (Active Comparator)
Started | 47 | 55
Completed | 41 | 47
Not Completed | 6 | 8
Not completed — Lost to Follow-up | 6 | 6
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Periodontal Intervention (Experimental) | Periodontal Prophylaxis (Active Comparator) | Total
Number analyzed (Participants) | 47 | 55 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (9.4) | 45.5 (8.1) | 45.5 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 30 | 54
  Male | 23 | 25 | 48
Race/Ethnicity, Customized [Number; unit: participants] — Ethnicity self reported by the participant of this clinical trial.
  participants
    White | 6 | 5 | 11
    Black | 5 | 5 | 10
    Indian | 0 | 3 | 3
    Mixed ethnicity | 36 | 42 | 78
Smoking status [Number; unit: participants]
  Currently smoking | 12 | 14 | 26
  Never smoker | 24 | 28 | 52
  Former smoker | 11 | 13 | 24
Formal education [Number; unit: participants]
  Elementary education (1 to 5 years) | 14 | 17 | 31
  Secondary education (6 to 11 years) | 22 | 25 | 47
  Higher education (12 or more years) | 11 | 13 | 24
Family monthly income [Number; unit: participants] — Economic incomes are presented in United States Dollars (USD). Exchange rate used in this study for the conversion of Colombian Pesos (COP) to USD: 2000 COP = 1 USD.
  participants
    Less than $300 USD | 19 | 23 | 42
    ≥ $300 and ≤ $600 USD | 24 | 22 | 46
    More than $600 USD | 4 | 10 | 14
Medical insurance [Number; unit: participants]
  None | 5 | 5 | 10
  State-subsidized healthcare | 30 | 34 | 64
  Contributory regime (private insurance) | 11 | 15 | 26
  Prepaid medicine plan | 1 | 1 | 2
Endothelium-dependent brachial artery flow-mediated dilatation [Mean (Standard Deviation); unit: Percentage of dilation] — Assessments of vascular function were performed in the morning, in a temperature controlled room, with participants required to fast for at least 8 hours.
  Flow-mediated endothelium dependent vasodilatation of the brachial artery (FMD) was determined using the technique previously described by Celermajer et al. (doi: 10.1016/0140-6736(92)93147-F.) and Coretti et al. ( doi: 10.1111/j.1399-302X.1996.tb00183.x.).
  FMD was calculated as the percentage of change in the diameter of brachial artery measured 45-60 s after cuff release in relation to the baseline measure.
  Percentage of dilation | 9.9 (7.4) | 9.9 (8.5) | 9.9 (7.9)
Serum C-reactive protein (CRP) [Mean (Standard Deviation); unit: mg/L] — Fasting plasma hs-CRP concentrations were determined using a solid-phase, chemiluminescent immunometric assay (Immulite 1000, Siemens). Baseline serum samples were not collected for one patient randomized into the periodontal prophylaxis group because of inaccessible veins.
  Number of patients analyzed:
  Periodontal intervention (n=47); Periodontal prophylaxis (n=54); Total (n=101).
  mg/L | 4 (7) | 3.1 (3.6) | 3.6 (5.4)

OUTCOME MEASURES:

1. Primary Outcome: Brachial Artery Flow-mediated Dilation
Description: All the assessments of vascular function were performed in the morning, in a temperature controlled room, with participants required to fast for at least 8 hours. Flow-mediated, endothelium dependent vasodilatation of the brachial artery (FMD) was measured using the technique described by Celermajer et al. using the guidelines reported by Coretti et al. FMD was calculated as the percentage of change in the diameter of brachial artery measured 45-60 s after cuff release in relation to the baseline measure (FMD%).
Time Frame: Baseline; 24 hours post periodontal therapy; 12 weeks post periodontal therapy
Population: The primary outcome (difference on endothelium-dependent brachial artery FMD at baseline and three months after randomization) and the secondary outcome (hs-CRP, glucose, blood lipid profile and cardiovascular biomarkers) were analyzed using kruskal-wallis and unpaired t test depending on the distribution of the variables.
Measure: Mean (Standard Deviation); unit: Percentage of dilatation of brachial art
Arm/Group | Periodontal Intervention (Experimental) | Periodontal Prophylaxis (Active Comparator)
Number analyzed (Participants) | 41 | 46
Percentage of dilatation of brachial art
  Baseline | 10.2 (7.3) | 10.3 (8.7)
  24 hours | 13.1 (9.5) | 8.1 (7.8)
  12 weeks | 11.2 (9.7) | 9.7 (8.5)
Statistical Analysis 1: Comparison: Periodontal Intervention (Experimental) vs Periodontal Prophylaxis (Active Comparator); Analyzed variable: Brachial Artery Flow-mediated Dilation (baseline). Note: data analysis of patients who completed the study protocol (n=86). Intention-to-treat analysis analysis was not used because its application for the evaluation of continuous data would imply imputing missing data for patients lost to follow-up. Mean and standard deviation of flow-mediated dilatation, including data from all patients randomized in this study, is reported in the field of baseline characteristics; Test type: Superiority or Other; p = 0.98, Kruskal-Wallis — A P value of 0.05 was used as a cut-off for statistical significance; Non-parametric test appropriate for the analysis of non-normally distributed data
Statistical Analysis 2: Comparison: Periodontal Intervention (Experimental) vs Periodontal Prophylaxis (Active Comparator); Analyzed variable: Brachial Artery Flow-mediated Dilation (24 hours); Test type: Superiority or Other; p = 0.005, Kruskal-Wallis — A P value of 0.05 was used as a cut-off for statistical significance; Non-parametric test appropriate for the analysis of non-normally distributed data
Statistical Analysis 3: Comparison: Periodontal Intervention (Experimental) vs Periodontal Prophylaxis (Active Comparator); Statistical analysis: Brachial Artery Flow-mediated Dilation (12 weeks). Intention-to-treat analysis was not used because input of values for patients lost at follow-up will artificially amplify the precision of outcome measures. Higgins JPT, Deeks JJ, Altman DG (editors). Chapter 16: Special topics in statistics. In: Higgins JPT, Green S (editors). Cochrane Handbook for Systematic Reviews of Interventions. Version 5.0.1. The Cochrane Collaboration, 2008. www.cochrane-handbook.org; Test type: Superiority or Other; p = 0.43, Kruskal-Wallis — A P value of 0.05 was used as a cut-off for statistical significance; Non-parametric test appropriate for the analysis of non-normally distributed data

2. Secondary Outcome: High-sensitivity C-Reactive Protein
Description: The fasting plasma hs-CRP concentrations was evaluated using a quantitative solid-phase, chemiluminescent immunometric assay (Immulite 1000, Siemens).
Time Frame: Baseline; 24 hours post periodontal therapy; 12 weeks post periodontal therapy
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Periodontal Intervention (Experimental) | Periodontal Prophylaxis (Active Comparator)
Number analyzed (Participants) | 38 | 46
mg/L
  Baseline | 4.2 (7.5) | 3.1 (3.7)
  24 hours | 4.9 (6.7) | 4.1 (4.6)
  12 weeks | 3.3 (4.9) | 3.2 (3.8)

3. Secondary Outcome: Total Cholesterol
Time Frame: Baseline; 24 hours post periodontal therapy; 12 weeks post periodontal therapy
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Periodontal Intervention (Experimental) | Periodontal Prophylaxis (Active Comparator)
Number analyzed (Participants) | 40 | 46
mg/dL
  Baseline | 197 (38.7) | 192.4 (33.8)
  24 hours | 195.4 (40.9) | 186.9 (42.8)
  12 weeks | 203.9 (35.6) | 200.6 (39.5)

4. Secondary Outcome: White Blood Cell Count
Time Frame: Baseline; 24 hours post periodontal therapy; 12 weeks post periodontal therapy
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Periodontal Intervention (Experimental) | Periodontal Prophylaxis (Active Comparator)
Number analyzed (Participants) | 40 | 46
cells/mm^3
  Baseline | 6937 (2986) | 6380 (1682)
  24 hours | 6198 (2601) | 6088 (2411)
  12 weeks | 5464 (3160) | 5382 (2963)

5. Secondary Outcome: Subgingival Microbiota
Description: Polymerase chain reaction (PCR) was used for detection of the three red-complex periodontal pathogens in periodontal pockets: Porphyromonas gingivalis (Pg), Treponema denticola (Td) and Tannerella forsythia (Tf).
Time Frame: 12 weeks post-periodontal therapy
Measure: Number; unit: participants
Arm/Group | Periodontal Intervention (Experimental) | Periodontal Prophylaxis (Active Comparator)
Number analyzed (Participants) | 39 | 44
participants
  Participants positive for Pg | 31 | 42
  Participants positive for Td | 31 | 38
  Participants positive for Tf | 34 | 40
  Participants positive for Pg, Tf and Td | 25 | 37

6. Secondary Outcome: LDL Cholesterol
Time Frame: Baseline; 24 hours post periodontal therapy; 12 weeks post periodontal therapy
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Periodontal Intervention (Experimental) | Periodontal Prophylaxis (Active Comparator)
Number analyzed (Participants) | 40 | 46
mg/dL
  Baseline | 113.1 (37.6) | 106.4 (32.8)
  24 hours | 111.3 (41.3) | 104.6 (33.9)
  12 weeks | 119.9 (38.8) | 109.5 (42.8)

7. Secondary Outcome: Endothelial Leukocyte Adhesion Molecule-1 (E-Selectin)
Description: Multiplexed immuno-cytometric assay for the simultaneous measurement of MMP-9, MPO, tPAI-1, E-Selectin, ICAM-1, and VCAM-1 in serum samples (Milliplex® MAP kit, Human Cardiovascular Disease Panel 1, Millipore®).
  Luminex® 200™ IS Total System and xPONENT software were used for data acquisition and analysis.
Time Frame: 12 weeks post periodontal therapy
Population: Explanation of missing data in the intervention group: Blood samples obtained from two patients randomized to the periodontal intervention group were not suitable for the Luminex analysis.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Periodontal Intervention (Experimental) | Periodontal Prophylaxis (Active Comparator)
Number analyzed (Participants) | 38 | 46
ng/ml | 44.8 (28.7) | 42.9 (22.2)

8. Secondary Outcome: Intercellular Adhesion Molecule 1 (ICAM-1)
Time Frame: 12 weeks post periodontal therapy
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Periodontal Intervention (Experimental) | Periodontal Prophylaxis (Active Comparator)
Number analyzed (Participants) | 38 | 46
ng/ml | 247.1 (196.7) | 235.4 (229.6)

9. Secondary Outcome: Vascular Cell Adhesion Molecule 1 (VCAM-1)
Time Frame: 12 weeks post periodontal therapy
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Periodontal Intervention (Experimental) | Periodontal Prophylaxis (Active Comparator)
Number analyzed (Participants) | 38 | 46
ng/ml | 1601.6 (372.4) | 1588.1 (412.3)

10. Secondary Outcome: Myeloperoxidase (MPO)
Time Frame: 12 weeks post periodontal therapy
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Periodontal Intervention (Experimental) | Periodontal Prophylaxis (Active Comparator)
Number analyzed (Participants) | 38 | 46
ng/ml | 62.6 (60.9) | 83.8 (140.4)

11. Secondary Outcome: Matrix Metalloproteinase-9 (MMP-9)
Time Frame: 12 weeks post periodontal therapy
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Periodontal Intervention (Experimental) | Periodontal Prophylaxis (Active Comparator)
Number analyzed (Participants) | 38 | 46
ng/ml | 103.4 (58.5) | 110.5 (68.2)

12. Secondary Outcome: Tissue Plasminogen Activator Inhibitor-1 (tPAI-1)
Time Frame: 12 weeks post periodontal therapy
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Periodontal Intervention (Experimental) | Periodontal Prophylaxis (Active Comparator)
Number analyzed (Participants) | 38 | 46
ng/ml | 116.1 (74.1) | 110.7 (66.4)

ADVERSE EVENTS:
Time Frame: One day after periodontal therapy
Description: Method for data collection: semi-structured interview and examination of periodontal tissues.
Arm/Group | Periodontal Intervention (Experimental) | Periodontal Prophylaxis (Active Comparator)
Serious Adverse Events (participants affected / at risk) | 0/47 | 1/55
Other Adverse Events (participants affected / at risk) | 47/47 | 31/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Periodontal Intervention (Experimental) (N=47) | Periodontal Prophylaxis (Active Comparator) (N=55)
Motor vehicle traffic accident (Social circumstances) | 0 (0) | 1 (1) — Death
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Periodontal Intervention (Experimental) (N=47) | Periodontal Prophylaxis (Active Comparator) (N=55)
Swelling (Surgical and medical procedures) | 47 | 28 — Visual examination of periodontal tissues 24 h after periodontal therapy.
Gingival erythema or bleeding (Surgical and medical procedures) | 46 | 24 — Visual examination and patient interview 24 h after therapy. These adverse effects are frequently reported together (erythema is frequently a sign of gingival bleeding).
Periodontal pain (low-intensity) (Surgical and medical procedures) | 36 | 18 — Pain intensity was assessed by patient interview 24 h after periodontal therapy.

LIMITATIONS AND CAVEATS:
1. Patient recruitment take more time that previously expected, 2. Longer time than expected for the standardization for laboratory techniques, 3. Changes of the study personnel during patient recruitment and laboratory analysis of biological samples

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No